CLINICAL TRIAL: NCT03943056
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single- and Multiple-Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of BIIB091, a Bruton's Tyrosine Kinase (BTK) Inhibitor, in Healthy Adult Participants
Brief Title: A Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of BIIB091, a Bruton's Tyrosine Kinase (BTK) Inhibitor, in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 257HV101
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — BIIB091

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Single Ascending Dose (SAD): Cohort 1A (Experimental): Participants will receive dose level 1 of BIIB091 or placebo, orally, while fasting on Day 1.
  Interventions: Drug: BIIB091; Drug: Placebo
- (SAD): Cohort 2A (Experimental): Participants will receive dose level 2 of BIIB091 or placebo, orally, while fasting on Day 1.
  Interventions: Drug: BIIB091; Drug: Placebo
- (SAD): Cohort 3A (Experimental): Participants will receive dose level 3 of BIIB091 or placebo, orally, while fasting on Day 1, then again following a 7 day washout and high-fat meal.
  Interventions: Drug: BIIB091; Drug: Placebo
- (SAD): Cohort 4A (Experimental): Participants will receive dose level 4 of BIIB091 or placebo, orally, while fasting on Day 1.
  Interventions: Drug: BIIB091; Drug: Placebo
- (SAD): Cohort 5A (Experimental): Participants will receive dose level 5 of BIIB091 or placebo, orally, while fasting on Day 1.
  Interventions: Drug: BIIB091; Drug: Placebo
- Multiple Ascending Dose (MAD): Cohort 1B (Experimental): Participants will receive dose level 1 of BIIB091 or placebo, orally, twice daily (BID) for 13 days, and a single dose on Day 14.
  Interventions: Drug: BIIB091; Drug: Placebo
- (MAD): Cohort 2B (Experimental): Participants will receive dose level 2 of BIIB091 or placebo, orally, BID for 13 days, and a single dose on Day 14.
  Interventions: Drug: BIIB091; Drug: Placebo
- (MAD): Cohort 3B (Experimental): Participants will receive dose level 3 of BIIB091 or placebo, orally, BID for 13 days, and a single dose on Day 14.
  Interventions: Drug: BIIB091; Drug: Placebo

INTERVENTIONS:
Drug: BIIB091 — Administered as specified in the treatment arm.
Drug: Placebo — Administered as specified in the treatment arm.

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple oral doses of BIIB091 in healthy participants.This study will also determine the effect of food on the single oral dose pharmacokinetic (PK).

DETAILED DESCRIPTION:
Initial protocol recruitment and follow up was completed by 10 Jan 2020 with an optional cohort intended for completion by April 2020. Subsequently, a decision was made not to progress this optional cohort in light of COVID-19 which has resulted in a delay in reporting the actual completion date.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with applicable participant privacy regulations.
* Have a body mass index between 18 and 30 kg/m2, inclusive.
* All male participants must practice highly effective methods of contraception and not donate sperm during the study and for at least 1 spermatogenic cycle (90 days) after administration of last dose of study treatment.
* All female participants of childbearing potential must practice highly effective methods of contraception and not donate eggs during the study and for at least 90 days after their last dose of study treatment.
* Must be in good health as by the Investigator, based on medical history and screening evaluations.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic,hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* History of severe allergic or anaphylactic reactions, or of any allergic reactions that in the opinion of the Investigator are likely to be exacerbated by any component of the study treatment.
* History of, or ongoing, malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell carcinomas and squamous cell carcinomas that have been completely excised and considered cured at least 12 months prior to Check-in).
* Current enrollment or plan to enroll in any other drug, biological, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days prior to Check-in, or 5 half-lives of the drug or therapy, whichever is longer.
* Breastfeeding, pregnant, or planning to become pregnant during study participation.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Day 9 for SAD Cohorts; Baseline up to Day 24 for MAD Cohorts
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death, in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event), however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.

SECONDARY OUTCOMES:
Area Under the Curve from Time 0 to the Time of the Last Measurable Concentration (AUClast) | Baseline and multiple timepoints up to Day 3 for SAD Cohorts; Baseline and multiple timepoints up to Day 16 for MAD Cohorts
Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf) | Baseline and multiple timepoints up to Day 3
Maximum Observed Concentration (Cmax) | Baseline and multiple timepoints up to Day 3 for SAD Cohorts; Baseline and multiple timepoints up to Day 14 for MAD Cohorts
Time to Reach Maximum Observed Concentration (Tmax) | Baseline and multiple timepoints up to Day 3 for SAD Cohorts; Baseline and multiple timepoints up to Day 14 for MAD Cohorts
Elimination Half-Life (t½) | Baseline and multiple timepoints up to Day 3 for SAD Cohorts; Baseline and multiple timepoints up to Day 16 for MAD Cohorts
Apparent Total Body Clearance (CL/F) | Baseline and multiple timepoints up to Day 3 for SAD Cohorts; Baseline and multiple timepoints up to Day 16 for MAD Cohorts
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) | Baseline and multiple timepoints up to Day 3 for SAD Cohorts; Baseline and multiple timepoints up to Day 16 for MAD Cohorts
Amount of BIIB091 Excreted in Urine per Sampling Interval (Aeu) | Baseline and multiple timepoints up to Day 3
Percentage of BIIB091 Excreted in Urine per Sampling Interval (%Feu) | Baseline and multiple timepoints up to Day 3
Renal clearance (CLr) | Baseline and multiple timepoints up to Day 3
Area Under the Concentration-Time Curve Within a Dosing Interval (AUCtau) | Baseline and multiple timepoints up to Day 16
Accumulation Ratio (R) | Baseline and multiple timepoints up to Day 16
Trough concentration (Ctrough) | Baseline and multiple timepoints up to Day 16

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/